CLINICAL TRIAL: NCT04270188
Title: Prospective Study of the Evolution of Symptoms After Anterior Sacrospinofixation by Autologous Tissues
Brief Title: Evolution of Symptoms After Anterior Sacrospinofixation by Autologous Tissues
Acronym: SANTAU
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0077; 2020-A00350-39 (Other: ID-RCB)
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: middle anterior prolapse ≥ II (POP-Q classification); anterior prolapse ≥ II (POP-Q classification)
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anterior sacrospinofixation with autologous tissue: patients with middle and / or anterior prolapse ≥ II in the POP-Q classification and for whom an intervention by anterior sacrospinofixation by autologous tissues is planned.
  Interventions: Other: evolution of patient symptoms

INTERVENTIONS:
Other: evolution of patient symptoms — evolution of symptoms on the PGI-I scale (score 1, 2, or 3) 2 months after surgery

SUMMARY:
Prolapse is a pathology that can cause pelvic, urinary or sexual functional disorders and impaired quality of life. Although the use of vaginal mesh is a commonly practiced technique to correct prolapse, in recent years health officials have pointed to the lack of adequate safety and tolerability assessments of these implants. Currently, surgeons are therefore moving towards techniques without implants. The standard vaginal technique for the treatment of uterine prolapse is sacrospinofixation according to Richter. This technique can be performed without an implant, using autologous tissue.

Functional discomfort of patients is the main problem linked to the presence of prolapse. However, no study has yet evaluated the feelings of patients following the use of this sacrospinofixation technique by autologous tissues by vaginal route, which led us to set up this study.

The hypothesis is that the technique of anterior sacrospinofixation by autologous tissues improves the symptoms experienced by patients with an mid-level and / or anterior genital prolapse.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* middle and / or anterior genital prolapse (hysterocele and / or cystocele) requiring surgical correction of stage ≥ II in the POP-Q classification
* patients wanting an intervention because of the discomfort caused by the prolapse
* intervention planned by anterior sacrospinofixation by autologous tissues
* person having expressed his non-opposition

Exclusion Criteria:

* prolapse of stage < II in the POP-Q classification, or prolapse without functional impairment
* disorders involving an unacceptable risk of postoperative complications sought after questioning of the patient (blood coagulation disorders, immune system disorders, progressive diseases, etc.)
* reduced mobility of the lower limbs (not allowing positioning for surgery)
* pregnancy or any pregnancy plan for the duration of the study
* active or latent infection
* inability to understand the information given
* person deprived of liberty, under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years old with middle and / or anterior prolapse ≥ II in the POP-Q classification and for whom an intervention by anterior sacrospinofixation by autologous tissues is planned.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-07-11 (Estimated); Study Completion 2025-07-11 (Estimated)

PRIMARY OUTCOMES:
improvement of symptoms | at Month 2
  percentage of patients with symptom change on the PGI-I scale (score 1, 2, or 3)

CONTACTS AND LOCATIONS:
Overall Officials: Géry LAMBLIN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France